CLINICAL TRIAL: NCT00611156
Title: Bioactive Food Ingredients and Energy Metabolism: The Effects of Ginger, Black Pepper, Horseradish and Mustard on Meal-Induced Thermogenesis and Fat Oxidation
Brief Title: Examination of the Effects of Four Different Spices on Energy Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: B228-IHE-2006-NTG
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2007-08

CONDITIONS: Healthy
Keywords: Thermogenesis; Meal-induced thermogenesis; energy expenditure; fat oxidation; bioactive ingredients; spices; ginger; horseradish; black pepper; mustard
MeSH Terms: interventions — ginger extract; black pepper oil; Amines

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental): Spice
  Interventions: Dietary Supplement: ginger
- B (Experimental): Spice
  Interventions: Dietary Supplement: black pepper
- C (Experimental): Spice
  Interventions: Dietary Supplement: horseradish
- D (Experimental): Spice
  Interventions: Dietary Supplement: mustard
- E (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: ginger — added to a brunch meal
  Arms: A
Dietary Supplement: black pepper — Added to a brunch meal
  Arms: B
Dietary Supplement: horseradish — Added to a brunch meal
  Arms: C
Dietary Supplement: mustard — Added to a brunch meal
  Arms: D
Dietary Supplement: placebo — Added to a bruch meal
  Arms: E

SUMMARY:
The objective of this study is to examine whether four different spices (ginger, black pepper, horseradish and mustard) are able to increase energy metabolism.

Since chili and other spices have been shown to increase energy expenditure compared to placebo, we expect that some or all of the four spices may actually increase energy expenditure - although not to a large degree.

DETAILED DESCRIPTION:
Several pungent food ingredients, such as chili,and also other bioactive food ingredients, e.g. green tea, have been shown to be able to increase energy expenditure and fat oxidation during the hours following a meal containing the bioactive ingredient. Furthermore, we will also look at the subjects own feelings of appetite and thereby examine whether the appetite is affected by the spicy food. We expect to see some small effects on these parameters.

ELIGIBILITY:
Inclusion Criteria:

* male
* healthy and not use medication (regularly)
* normal weight
* non smoker
* tolerate and like spicy food
* stable body weight last two months

Exclusion Criteria:

* increased blood pressure
* abnormal EKG
* mental, metabolic and chronic diseases

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2006-10; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
energy expenditure | November 2007

SECONDARY OUTCOMES:
blood pressure | December 2007
heart rate | December 2007
VAS-scores for appetite, hunger, fullness, etc. - and palatability | November 2007
tolerance | November 2007
Fat and carbohydrate oxidation | November 2007
Meal-induced thermogenesis | November 2007

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor MD, Study Chair — Department of Human Nutrition, RVAU
Locations (1):
- Department of Human Nutrition, The Royal Veterinary and Agricultural University, Frederiksberg, Denmark

REFERENCES:
- [Derived] Gregersen NT, Belza A, Jensen MG, Ritz C, Bitz C, Hels O, Frandsen E, Mela DJ, Astrup A. Acute effects of mustard, horseradish, black pepper and ginger on energy expenditure, appetite, ad libitum energy intake and energy balance in human subjects. Br J Nutr. 2013 Feb 14;109(3):556-63. doi: 10.1017/S0007114512001201. Epub 2012 Jul 5. PMID 23021155